CLINICAL TRIAL: NCT03696576
Title: EMST And PhoRTE Training For Elderly Patients With Vocal Fold Atrophy
Brief Title: Expiratory Muscle Strength Training and Phonation Resistance Training Exercises For Elderly Patients With Vocal Fold Atrophy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the pandemic, recruitment ended earlier than expected and changes were required to alter data collection methods (and were approved by the IRB). Additional changes were also made to the protocol to move the study to an online platform.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Amanda Gillespie, Assitant professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00109224; PRO18040682 (Other: University of Pittsburgh)
Record Dates: First submitted 2018-09-20; First posted 2018-10-04 (Actual); Results first posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Voice Disorder; Vocal Cord Atrophy; Presbyphonia
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Speech Language Pathologists (SLPs) will not know which group the participants have been randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PhoRTE (Active Comparator): This group will undergo standard PhoRTE therapy.
  Interventions: Behavioral: PhoRTE
- PhoRTE + EMST (Experimental): This group will undergo standard PhoRTE therapy with the addition of expiratory muscle strength training using the EMST device.
  Interventions: Device: EMST; Behavioral: PhoRTE

INTERVENTIONS:
Device: EMST — Training of the respiratory system muscles using the EMST device.
  Arms: PhoRTE + EMST
Behavioral: PhoRTE — Completing of PhoRTE voice therapy.

SUMMARY:
The larynx and vocal folds undergo many age-related changes in their physiology and structure that can lead to undesirable effects on the voice, with changes in the respiratory system compounding these deficits. These changes, also called presbyphonia, can have serious detrimental effects on the lives of elderly individuals. There are few studies that have evaluated the use of voice therapy treatment options for these patients. The primary aim of this study is to test whether the addition of expiratory muscle strength training (EMST) to a current, validated voice therapy protocol aimed at treating presbyphonia, (phonation resistance training, PhoRTE) can improve outcomes of therapy.

DETAILED DESCRIPTION:
The purpose of this study is to test whether the addition of EMST to PhoRTE Voice Therapy is at least as effective as PhoRTE alone for improving acoustic, aerodynamic, and patient-reported outcomes in patients affected by age-related vocal fold atrophy.

Voice therapy is often the first-line treatment for patients experiencing presbyphonia. Despite being the most common treatment for presbyphonia, scant literature exists on the efficacy of voice therapy for these patients. The current proposal aims to add to this growing body of literature. In general, studies of existing voice therapy programs for presbyphonia have demonstrated success in achieving improvement in aerodynamic (increased subglottal pressure), acoustic (increased shimmer, jitter, and decreased noise-to-harmonics ratio), and patient-centered outcomes (reduction in Voice Handicap Index scores, decreased phonatory effort). Ziegler et al. conducted a study comparing a standard voice therapy, Vocal Function Exercises (VFE) and Phonation Resistance Training Exercises (PhoRTE) and found that both therapies improved outcomes of voice-related quality of life, but only PhoRTE gave a statistically significant reduction in perceived phonatory effort. A specific therapy designed to address age-related changes to respiratory system is expiratory muscle strength training (EMST). EMST devices are loaded with a resistive spring which opens when a desired level of expiratory pressure is reached and maintained. Maintenance of consistent subglottal pressure is the foundation for phonation. EMST device training improves active expiratory muscle forces required for high-pressure activities such as long utterances or loud speech in vocally healthy individuals. When used in conjunction with traditional voice therapy, EMST use has also shown to increase maximum phonation time, maximum expiratory pressure, dynamic range, subglottal pressure, and perception of voice handicap in professional voice users over traditional voice therapy alone. The theoretical underpinnings for treatment of vocal fold atrophy with EMST are clear, as it addresses many of the common goals of treatment in patients with presbyphonia, but it has not yet been tested as a possible adjunctive treatment for patients undergoing voice therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* Diagnosis of presbyphonia (vocal fold atrophy) made by a fellowship-trained laryngologist and a voice specialized speech language pathologist
* Willingness to be randomized to one of two treatments

Exclusion Criteria:

* Any concomitant laryngeal diagnoses or diseases known to affect voice function, including: amyloidosis, arytenoid dislocation, laryngeal cancer, cricoarytenoid fixation, vocal fold cyst(s), vocal nodules, vocal fold polyp(s), dysplasia, vocal fold fibrous mass(es), glottal web, vocal fold immobility, laryngeal stenosis, laryngocele, leukoplakia, Parkinson's disease, Reinke's edema, respiratory recurrent pneumonia, sarcoidosis, spasmodic dysphonia
* Any chronic lower airway disease such as chronic obstructive pulmonary disease (COPD), asthma, chronic bronchitis, emphysema, cystic fibrosis
* History of acute stroke
* Untreated hypertension
* Untreated gastroesophageal reflux disease (GERD)

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Gillespie, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - University of Pittsburgh Voice Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
only de-identified data will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: during and through data analysis
Access Criteria: additional researchers may receive de-identified information only if a data use agreement has been executed.

REFERENCES:
- [Background] Kost K, Parham K. Presbyphonia: What can be done? Ear Nose Throat J. 2017 Mar;96(3):108-110. doi: 10.1177/014556131709600309. No abstract available. PMID 28346640
- [Background] Polkey MI, Harris ML, Hughes PD, Hamnegard CH, Lyons D, Green M, Moxham J. The contractile properties of the elderly human diaphragm. Am J Respir Crit Care Med. 1997 May;155(5):1560-4. doi: 10.1164/ajrccm.155.5.9154857.
- [Background] Janssens JP, Pache JC, Nicod LP. Physiological changes in respiratory function associated with ageing. Eur Respir J. 1999 Jan;13(1):197-205. doi: 10.1034/j.1399-3003.1999.13a36.x. PMID 10836348
- [Background] Skloot GS. The Effects of Aging on Lung Structure and Function. Clin Geriatr Med. 2017 Nov;33(4):447-457. doi: 10.1016/j.cger.2017.06.001. Epub 2017 Aug 19. PMID 28991643
- [Background] Thomas LB, Harrison AL, Stemple JC. Aging thyroarytenoid and limb skeletal muscle: lessons in contrast. J Voice. 2008 Jul;22(4):430-50. doi: 10.1016/j.jvoice.2006.11.006. Epub 2007 Jan 22. PMID 17241767
- [Background] Takano S, Kimura M, Nito T, Imagawa H, Sakakibara K, Tayama N. Clinical analysis of presbylarynx--vocal fold atrophy in elderly individuals. Auris Nasus Larynx. 2010 Aug;37(4):461-4. doi: 10.1016/j.anl.2009.11.013. Epub 2009 Dec 28. PMID 20036792
- [Background] Davids T, Klein AM, Johns MM 3rd. Current dysphonia trends in patients over the age of 65: is vocal atrophy becoming more prevalent? Laryngoscope. 2012 Feb;122(2):332-5. doi: 10.1002/lary.22397. Epub 2012 Jan 17. PMID 22252988
- [Background] Roy N, Stemple J, Merrill RM, Thomas L. Epidemiology of voice disorders in the elderly: preliminary findings. Laryngoscope. 2007 Apr;117(4):628-33. doi: 10.1097/MLG.0b013e3180306da1. PMID 17429872
- [Background] Golub JS, Chen PH, Otto KJ, Hapner E, Johns MM 3rd. Prevalence of perceived dysphonia in a geriatric population. J Am Geriatr Soc. 2006 Nov;54(11):1736-9. doi: 10.1111/j.1532-5415.2006.00915.x. PMID 17087701
- [Background] Gregory ND, Chandran S, Lurie D, Sataloff RT. Voice disorders in the elderly. J Voice. 2012 Mar;26(2):254-8. doi: 10.1016/j.jvoice.2010.10.024. Epub 2011 May 6. PMID 21530163
- [Background] Palmer AD, Newsom JT, Rook KS. How does difficulty communicating affect the social relationships of older adults? An exploration using data from a national survey. J Commun Disord. 2016 Jul-Aug;62:131-46. doi: 10.1016/j.jcomdis.2016.06.002. Epub 2016 Jun 22. PMID 27420152
- [Background] Holt-Lunstad J, Smith TB, Layton JB. Social relationships and mortality risk: a meta-analytic review. PLoS Med. 2010 Jul 27;7(7):e1000316. doi: 10.1371/journal.pmed.1000316. PMID 20668659
- [Background] Marmor S, Horvath KJ, Lim KO, Misono S. Voice problems and depression among adults in the United States. Laryngoscope. 2016 Aug;126(8):1859-64. doi: 10.1002/lary.25819. Epub 2015 Dec 21. PMID 26691195
- [Background] Tay EY, Phyland DJ, Oates J. The effect of vocal function exercises on the voices of aging community choral singers. J Voice. 2012 Sep;26(5):672.e19-27. doi: 10.1016/j.jvoice.2011.12.014. Epub 2012 Jun 19. PMID 22717496
- [Background] Gorman S, Weinrich B, Lee L, Stemple JC. Aerodynamic changes as a result of vocal function exercises in elderly men. Laryngoscope. 2008 Oct;118(10):1900-3. doi: 10.1097/MLG.0b013e31817f9822. PMID 18622308
- [Background] Ziegler A, Verdolini Abbott K, Johns M, Klein A, Hapner ER. Preliminary data on two voice therapy interventions in the treatment of presbyphonia. Laryngoscope. 2014 Aug;124(8):1869-76. doi: 10.1002/lary.24548. Epub 2014 Jan 29. PMID 24375313
- [Background] Caskey CI, Zerhouni EA, Fishman EK, Rahmouni AD. Aging of the diaphragm: a CT study. Radiology. 1989 May;171(2):385-9. doi: 10.1148/radiology.171.2.2704802.
- [Background] Kim J, Sapienza CM. Implications of expiratory muscle strength training for rehabilitation of the elderly: Tutorial. J Rehabil Res Dev. 2005 Mar-Apr;42(2):211-24. doi: 10.1682/jrrd.2004.07.0077. PMID 15944886
- [Background] Enright PL, Kronmal RA, Higgins MW, Schenker MB, Haponik EF. Prevalence and correlates of respiratory symptoms and disease in the elderly. Cardiovascular Health Study. Chest. 1994 Sep;106(3):827-34. doi: 10.1378/chest.106.3.827. PMID 8082366
- [Background] Nam DH, Lim JY, Ahn CM, Choi HS. Specially programmed respiratory muscle training for singers by using respiratory muscle training device (Ultrabreathe). Yonsei Med J. 2004 Oct 31;45(5):810-7. doi: 10.3349/ymj.2004.45.5.810. PMID 15515190
- [Background] Wingate JM, Brown WS, Shrivastav R, Davenport P, Sapienza CM. Treatment outcomes for professional voice users. J Voice. 2007 Jul;21(4):433-49. doi: 10.1016/j.jvoice.2006.01.001. Epub 2006 Apr 3. PMID 16581229
- [Background] Baker S, Davenport P, Sapienza C. Examination of strength training and detraining effects in expiratory muscles. J Speech Lang Hear Res. 2005 Dec;48(6):1325-33. doi: 10.1044/1092-4388(2005/092). PMID 16478374
- [Background] Sapienza CM, Wheeler K. Respiratory muscle strength training: functional outcomes versus plasticity. Semin Speech Lang. 2006 Nov;27(4):236-44. doi: 10.1055/s-2006-955114. PMID 17117350
- [Background] Murry T. Subglottal pressure and airflow measures during vocal fry phonation. J Speech Hear Res. 1971 Sep;14(3):544-51. doi: 10.1044/jshr.1403.544. No abstract available. PMID 5163888
- [Background] Smitheran JR, Hixon TJ. A clinical method for estimating laryngeal airway resistance during vowel production. J Speech Hear Disord. 1981 May;46(2):138-46. doi: 10.1044/jshd.4602.138. PMID 7253590
- [Background] Laciuga H, Rosenbek JC, Davenport PW, Sapienza CM. Functional outcomes associated with expiratory muscle strength training: narrative review. J Rehabil Res Dev. 2014;51(4):535-46. doi: 10.1682/JRRD.2013.03.0076. PMID 25144167
- [Background] Rosen CA, Lee AS, Osborne J, Zullo T, Murry T. Development and validation of the voice handicap index-10. Laryngoscope. 2004 Sep;114(9):1549-56. doi: 10.1097/00005537-200409000-00009. PMID 15475780
- [Background] Gillespie AI, Dastolfo C, Magid N, Gartner-Schmidt J. Acoustic analysis of four common voice diagnoses: moving toward disorder-specific assessment. J Voice. 2014 Sep;28(5):582-8. doi: 10.1016/j.jvoice.2014.02.002. Epub 2014 May 28. PMID 24880672
- [Background] Awan SN, Roy N, Jette ME, Meltzner GS, Hillman RE. Quantifying dysphonia severity using a spectral/cepstral-based acoustic index: Comparisons with auditory-perceptual judgements from the CAPE-V. Clin Linguist Phon. 2010 Sep;24(9):742-58. doi: 10.3109/02699206.2010.492446. PMID 20687828
- [Background] Kempster GB, Gerratt BR, Verdolini Abbott K, Barkmeier-Kraemer J, Hillman RE. Consensus auditory-perceptual evaluation of voice: development of a standardized clinical protocol. Am J Speech Lang Pathol. 2009 May;18(2):124-32. doi: 10.1044/1058-0360(2008/08-0017). Epub 2008 Oct 16. PMID 18930908
- [Background] Etter NM, Hapner ER, Barkmeier-Kraemer JM, Gartner-Schmidt JL, Dressler EV, Stemple JC. Aging Voice Index (AVI): Reliability and Validity of a Voice Quality of Life Scale for Older Adults. J Voice. 2019 Sep;33(5):807.e7-807.e12. doi: 10.1016/j.jvoice.2018.04.006. Epub 2018 May 7. PMID 29748025
- [Background] Gartner-Schmidt J, Rosen C. Treatment success for age-related vocal fold atrophy. Laryngoscope. 2011 Mar;121(3):585-9. doi: 10.1002/lary.21122. Epub 2010 Aug 3. PMID 21344441
- [Background] Sauder C, Roy N, Tanner K, Houtz DR, Smith ME. Vocal function exercises for presbylaryngis: a multidimensional assessment of treatment outcomes. Ann Otol Rhinol Laryngol. 2010 Jul;119(7):460-7. doi: 10.1177/000348941011900706. PMID 20734967
- [Background] Fairbanks G. Voice and articulation drill book. 2nd ed. New York: Harper and Row; 1960.
- [Background] Statistics FIFoAR. Older Americans 2010: Key Indicators of Well-Being. US Government Printing Office. 2010.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited for the study from September 2018 until March 2020.
Period: Overall Study
Arm/Group | PhoRTE | PhoRTE + EMST
Started | 13 | 11
Completed | 10 | 6
Not Completed | 3 | 5
Not completed — Soreness of throat after therapy | 1 | 1
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PhoRTE | PhoRTE + EMST | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.10 (7.91) | 75.22 (8.12) | 73.53 (7.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 8 | 7 | 15
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Voice Handicap Index-10 (VHI-10) Score
Description: The Voice Handicap Index-10 (VHI-10) is a validated assessment instrument that quantifies patient perceptions of his or her own voice handicap. A lower score on the VHI-10 indicates perception of a lesser voice handicap than a high score. Scores range from 0 to 40.
Time Frame: At each study visit through study completion; Time 0 (therapy visit 1-Baseline), follow-up week 1 (therapy visit 2), follow-up week 2 (therapy visit 3),follow-up week 3 (therapy visit 4), follow-up week 5 (follow up visit)
Population: Number of participants analyzed is different in each time point, due to difficulties bringing participants into the clinic because of COVID-19.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- PhoRTE: This group received standard PhoRTE therapy.
  PhoRTE: Completing of PhoRTE voice therapy.
- PhoRTE + EMST: This group received standard PhoRTE therapy with the addition of expiratory muscle strength training using the EMST device.
  EMST: Training of the respiratory system muscles using the EMST device.
  PhoRTE: Completing of PhoRTE voice therapy.
Arm/Group | PhoRTE | PhoRTE + EMST
Number analyzed (Participants) | 13 | 11
score on a scale
  Baseline: number analyzed (Participants) | 10 | 11
  Baseline | 15.80 (6.94) | 17.45 (8.55)
  Follow up-week 1 | 18.85 (9.5) | 20.54 (10.53)
  Follow up-week 2: number analyzed (Participants) | 12 | 9
  Follow up-week 2 | 17.00 (9.86) | 17.00 (12.22)
  Follow up-week 3: number analyzed (Participants) | 11 | 6
  Follow up-week 3 | 14.09 (9.76) | 15.67 (11.94)
  Follow up-week 4: number analyzed (Participants) | 10 | 6
  Follow up-week 4 | 12.00 (11.07) | 10.17 (6.97)
  Follow up-week 5: number analyzed (Participants) | 10 | 6
  Follow up-week 5 | 13.3 (10.86) | 10.50 (9.69)

2. Secondary Outcome: AVI Score at Baseline and Follow up (5 Weeks)
Description: The Aging Voice Index (AVI) is a validated instrument that measures quality of life in older adults with voice disorders. A higher score indicates worse quality of life. Scores range from 0 to 92.
Time Frame: At initial therapy visit (Baseline) and final follow up-visit (Follow up - week 5)
Population: All participants were assessed for this outcome measure. 13 participants in the PhoRTE arm and 11 participants in the PhoRTE + EMST arm at baseline and follow up.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PhoRTE | PhoRTE + EMST
Number analyzed (Participants) | 13 | 11
score on a scale
  Baseline | 41.54 (6.19) | 43.64 (6.73)
  Follow Up | 23.13 (6.72) | 27.36 (8.23)

3. Secondary Outcome: Maximum Expiratory Pressure (MEP)
Description: Maximum Expiratory Pressure (MEP) was measured using a handheld manometer (Micro Direct Respiratory Pressure Meter, MicroRPM, Med-Electronics, Beltsville, MD, United States) at baseline and after 5 weeks of therapy. Participants were instructed to blow with maximum force into the MicroRPM device over 10 trials, and the participant's best three trials were used to calculate their average MEP.
Time Frame: At initial therapy visit (Baseline) and final follow up-visit (week 5)
Measure: Mean (Standard Error); unit: cm H2O
Arm/Group | PhoRTE | PhoRTE + EMST
Number analyzed (Participants) | 13 | 11
cm H2O
  Baseline | 43.08 (7.85) | 49.18 (8.20)
  Follow Up | 51.32 (8.83) | 81.81 (9.94)

4. Secondary Outcome: Phonatory Airflow in Speech at Baseline and 5 Weeks
Description: Aerodynamic measures were collected and analyzed via the Phonatory Aerodynamic System 6600 (PAS; PENTAX Medical, Montvale, NJ, United States) using the first four sentences of the Rainbow Passage. Aerodynamic measures included mean airflow during voicing and number of breaths taken. The PAS captured phonatory aerodynamic functioning using a pneumotach coupled to a facemask, with external microphone. During speech, expired air flows through the pneumotach, which consists of a stainless-steel mesh screen with pressure transducers on either side. The system calculates the pressure difference across the screen to determine airflow rate. The microphone is positioned at the end of the pneumotach and internally calibrated per system specifications to represent a mouth-to-microphone distance of 15 cm. The participant sat with the facemask held snugly over their nose and mouth while they read the first fou
Time Frame: At initial therapy visit (Baseline) and final follow up-visit (week 5)
Measure: Mean (Standard Error); unit: Liters/second
Arm/Group | PhoRTE | PhoRTE + EMST
Number analyzed (Participants) | 13 | 11
Liters/second
  Baseline | 0.29 (0.05) | 0.18 (0.06)
  Follow Up | 0.13 (0.07) | 0.12 (0.08)

5. Secondary Outcome: Number of Breaths at Baseline and Follow up (5 Weeks)
Description: Aerodynamic measurement: mean number of breaths in reading of a standard passage (The Rainbow Passage).
Time Frame: At initial therapy visit (Baseline) and final follow up-visit (week 5)
Measure: Mean (Standard Error); unit: number of breaths
Arm/Group | PhoRTE | PhoRTE + EMST
Number analyzed (Participants) | 13 | 11
number of breaths
  Baseline | 7.17 (0.96) | 6.59 (1.13)
  Follow Up | 7.36 (1) | 5.52 (1.29)

6. Secondary Outcome: Mean Cepstral Spectral Index of Dysphonia (CSID) Measurements While Reading Functional Phrases at Baseline and 5 Weeks
Description: Cepstral Spectral Index of Dysphonia (CSID) is a multifactorial estimate of dysphonia severity that correlates with an auditory perceptual rating of overall voice severity using a 0-100 visual analog scale. Components of the algorithm include the cepstral peak prominence and its standard deviation, the low to high spectral ratio and its standard deviation. Typically, CSID limits are 0-100, but very severe voices may exceed 100, and very periodic, normal voices may be less than 0.
Time Frame: Baseline (At initial therapy visit) and final follow up-visit (week 5)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PhoRTE | PhoRTE + EMST
Number analyzed (Participants) | 13 | 11
score on a scale
  Baseline | 26.05 (7.15) | 28.85 (7.84)
  Follow Up | 12.08 (8.57) | 20.7 (9.94)

7. Secondary Outcome: Cepstral Spectral Index of Dysphonia (CSID) Measurements at Baseline and 5 Weeks
Description: as for outcome 6
Time Frame: Baseline (At initial therapy visit) and final follow up-visit (week 5)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PhoRTE | PhoRTE + EMST
Number analyzed (Participants) | 13 | 11
score on a scale
  Baseline | 33.93 (8.02) | 42.9 (8.79)
  Follow Up | 13.08 (10.39) | 41.56 (12.27)

8. Secondary Outcome: Duration of Standard Reading Passage at Baseline and Follow up (5 Weeks)
Description: Aerodynamic measurement; mean duration to complete the reading of a standard passage (The Rainbow Passage).
Time Frame: At initial therapy visit (Baseline) and final follow up-visit (week 5)
Measure: Mean (Standard Error); unit: seconds
Arm/Group | PhoRTE | PhoRTE + EMST
Number analyzed (Participants) | 13 | 11
seconds
  Baseline | 27.23 (1.54) | 28.56 (1.61)
  Follow up | 25.31 (1.84) | 24.93 (2.11)

9. Secondary Outcome: Cepstral Peak Prominence at Baseline and 5 Weeks Follow up
Description: Acoustic measurement: Cepstral Peak Prominence and its standard deviation while reading functional phrases.
Time Frame: At initial therapy visit (Baseline) and final follow up-visit (after week 5)
Measure: Mean (Standard Error); unit: dB
Arm/Group | PhoRTE | PhoRTE + EMST
Number analyzed (Participants) | 13 | 11
dB
  Baseline | 8.05 (0.98) | 7.13 (1.07)
  Follow Up | 11.32 (1.27) | 7.68 (1.50)

10. Secondary Outcome: Cepstral Peak Prominence (CPP) Fundamental Frequency (F0) at Baseline and Follow up (5 Weeks)
Description: Acoustic measurement: CPP F0 while reading functional phrases.
Time Frame: At initial therapy visit (Baseline) and final follow up-visit (week 5)
Measure: Mean (Standard Error); unit: Hz
Arm/Group | PhoRTE | PhoRTE + EMST
Number analyzed (Participants) | 13 | 11
Hz
  Baseline | 166.21 (14.51) | 167.04 (15.9)
  Follow Up | 160.97 (15.81) | 178.09 (17.86)

11. Secondary Outcome: Mean Fundamental Frequency in Sentence at Baseline and at 5 Weeks
Description: Aerodynamic measurement: mean F0 in reading of a standard passage (The Rainbow Passage).
Time Frame: At initial therapy visit (Baseline) and final follow up-visit (week 5)
Population: All participants were assessed for this outcome measure. 13 participants in the PhoRTE arm and 11 participants in the PhoRTE + EMST arm, at baseline and follow up.
Measure: Mean (Standard Error); unit: Hz
Arm/Group | PhoRTE | PhoRTE + EMST
Number analyzed (Participants) | 13 | 11
Hz
  Baseline | 166.31 (8.66) | 152.78 (9.04)
  Follow Up | 177.09 (10.15) | 156.81 (11.55)

12. Secondary Outcome: Vocal Intensity at Baseline and Follow up
Description: Acoustic measurement: mean vocal intensity in dB SPL while reading functional phrases.
Time Frame: At initial therapy visit (baseline) and final follow up-visit (week 5)
Population: as for outcome 11
Measure: Mean (Standard Error); unit: dB SPL
Arm/Group | PhoRTE | PhoRTE + EMST
Number analyzed (Participants) | 13 | 11
dB SPL
  Baseline | 74.22 (1.49) | 76.48 (1.56)
  Follow Up | 78.06 (1.95) | 73.56 (2.31)

13. Secondary Outcome: Mean Change In Overall Voice Severity at 5 Weeks
Description: Overall voice severity determined by Consensus Auditory Perceptual Evaluation - Voice (CAPE-V) score provided by blinded raters. The visual analog scale for overall voice severity used. Minimum score = 0, Maximum score = 100. Higher values indicate worse voice.
Time Frame: At initial therapy visit and final follow up-visit, after week 5
Population: Auditory perceptual measurements of overall voice severity were not collected, thus not analyzed, due to having to convert to tele-health due to COVID-19 pandemic.
Arm/Group | PhoRTE | PhoRTE + EMST
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | PhoRTE | PhoRTE + EMST
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT03696576/Prot_SAP_000.pdf